CLINICAL TRIAL: NCT05082844
Title: Evaluation of Mid- to Long-term Clinical and Radiological Outcomes of Surgical Treatment for Rotator Cuff Injury in Patients Over 70
Brief Title: Evaluation of Clinical and Radiographic Outcomes of Surgical Treatment for Rotator Cuff Injury in Patients Over 70
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Institutional research funds needed to perform imaging examinations under the study protocol have expired due to organizational issues
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUFF70
Record Dates: First submitted 2021-08-09; First posted 2021-10-19 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2022-09

CONDITIONS: Cuff Rotator Syndrome
Keywords: cuff rotator; retrospective study; prospective study; long-term clinical evaluation; long-term radiological evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of clinical and radiographic findings after surgical treatment for cuff rotator lesion (Experimental): Evaluation of the clinical-radiological results from the case series of patients surgically treated for cuff rotator lesions from 2009 to 2020 at the Shoulder-Elbow Department . At 12 months the result is considered stabilized, so we will proceed to collect all case histories that have passed this follow-up period.
  Interventions: Radiation: MRI assessment

INTERVENTIONS:
Radiation: MRI assessment — Evaluation of the clinical-radiological results from the case series of patients surgically treated for cuff rotator lesions from 2009 to 2020 at the Shoulder-Elbow Department . At 12 months the result is considered stabilized, so we will proceed to collect all case histories that have passed this follow-up period.

SUMMARY:
The aim of the study is to document the clinical-radiological results from the case series of patients surgically treated for rotator cuff lesions from 2009 to 2020 at the Rizzoli Orthopaedic Institute Shoulder-Elbow Department.

DETAILED DESCRIPTION:
110 patients surgically treated for rotator cuff lesions from 2009 to 2020 will be included in a retrospective-prospective and interventional study with clinical and radiological evaluation at follow-up of at least 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. ≥70 years of age at the time of rotator cuff repair surgery
2. Males and Females
3. Patients surgically treated for rotator cuff injury between 2009 and 2020 at the Shoulder-Elbow Department of the Rizzoli Orthopaedic Institute

Exclusion Criteria:

* All available patients will be invited to undergo clinical examination and radiological examination. In case some patients cannot undergo MRI due to possible contraindications, they will still be seen to collect the primary clinical outcome

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Constant score | At least 12 months after cuff rotator lesion surgery
  The constant score is the most commonly used questionnaire for evaluating treatment outcomes of shoulder disorders. It's the scoring system recommended by the European Society of Shoulder and Elbow Surgery (SECEC / ESSE). It has the advantages of including pain score, functional assessment, range of motion, and strength measures. A high score corresponds to a great quality of function

SECONDARY OUTCOMES:
Visual Analog Scale (VAS): | At least 12 months after cuff rotator lesion surgery
  Analogue scale represented by a line of 10 cm length, ranging from "absence of pain" to "the worst imaginable pain "
Simple Shoulder Test (SST) | At least at leat 12 months after cuff rotator lesion surgery
  SST test consists of 12 questions about physical functioning with dichotomous response options (yes or no). Scores range from 0 (worst) to 100 (best) and are reported as the percentage of items answered in the affirmative by the patient
Short Form-12 (SF-12): | At least 12 months after cuff rotator lesion surgery
  SF-12 serves as a generic indicator of quality of life and assesses the individual's subjective perception of health, understood as biopsychosocial well-being. Through 12 of the 36 questions of the original questionnaire, the SF-12 investigates 8 different aspects related to health status: physical activity, role limitations due to physical health, emotional state, physical pain, perception of general health status, vitality, social activities and mental health; the synthesis of the total scores allows to build two synthetic indices, a physical health index (PCS-12) and a mental health index (MCS-12). The lower the score of the two indices, indicatively below 20 points, the greater the level of disability.
Treatment opinion post- surgery | At least 12 months after cuff rotator lesion surgery
  Patient satisfaction with their post-surgery recovery status will be assessed.
Magnetic Resonance Imaging | At least 12 months after cuff rotator lesion surgery
  Magnetic Resonace Imaging will be carried for evaluating a possible plica retraction.

REFERENCES:
- [Background] Longo UG, Margiotti K, Petrillo S, Rizzello G, Fusilli C, Maffulli N, De Luca A, Denaro V. Genetics of rotator cuff tears: no association of col5a1 gene in a case-control study. BMC Med Genet. 2018 Dec 20;19(1):217. doi: 10.1186/s12881-018-0727-1. PMID 30572822
- [Background] Hattrup SJ. Rotator cuff repair: relevance of patient age. J Shoulder Elbow Surg. 1995 Mar-Apr;4(2):95-100. doi: 10.1016/s1058-2746(05)80061-8. PMID 7600171
- [Background] Merolla G, Paladini P, Saporito M, Porcellini G. Conservative management of rotator cuff tears: literature review and proposal for a prognostic. Prediction Score. Muscles Ligaments Tendons J. 2011 Oct 30;1(1):12-9. Print 2011 Jan. PMID 23738239
- [Background] Yamaguchi K. Mini-open rotator cuff repair: an updated perspective. Instr Course Lect. 2001;50:53-61. PMID 11372355
- [Background] Robinson PM, Wilson J, Dalal S, Parker RA, Norburn P, Roy BR. Rotator cuff repair in patients over 70 years of age: early outcomes and risk factors associated with re-tear. Bone Joint J. 2013 Feb;95-B(2):199-205. doi: 10.1302/0301-620X.95B2.30246. PMID 23365029
- [Background] Geary MB, Elfar JC. Rotator Cuff Tears in the Elderly Patients. Geriatr Orthop Surg Rehabil. 2015 Sep;6(3):220-4. doi: 10.1177/2151458515583895. PMID 26328240
- [Background] Charousset C, Bellaiche L, Kalra K, Petrover D. Arthroscopic repair of full-thickness rotator cuff tears: is there tendon healing in patients aged 65 years or older? Arthroscopy. 2010 Mar;26(3):302-9. doi: 10.1016/j.arthro.2009.08.027. PMID 20206038
- [Background] Bhatia S, Greenspoon JA, Horan MP, Warth RJ, Millett PJ. Two-Year Outcomes After Arthroscopic Rotator Cuff Repair in Recreational Athletes Older Than 70 Years. Am J Sports Med. 2015 Jul;43(7):1737-42. doi: 10.1177/0363546515577623. Epub 2015 Apr 1. PMID 25834140